CLINICAL TRIAL: NCT06449859
Title: A Phase I Clinical Trial to Evaluate the Safety, Tolerability, and Pharmacokinetic Profile of TQC2938 Injection in Healthy Adult Subjects After Single and Multiple Administration
Brief Title: A Clinical Trial of TQC2938 Injection in Healthy Adult Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQC2938-I-01
Record Dates: First submitted 2024-06-03; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- TQC2938 Injection (52.5mg/0.35ml) (Experimental): TQC2938 Injection is administered as a single dose of subcutaneous (SC) injection.
  Interventions: Drug: TQC2938 Injection
- TQC2938 Injection (210mg/1.4ml)-subcutaneous injection (Experimental): TQC2938 Injection is administered as a single dose of subcutaneous injection.
  Interventions: Drug: TQC2938 Injection
- TQC2938 Injection (210mg/1.4ml)-intravenous injection (Experimental): TQC2938 Injection is administered as a single dose of intravenous (IV) injection .
  Interventions: Drug: TQC2938 Injection
- TQC2938 Injection (420mg/2.8ml) (Experimental): TQC2938 Injection is administered as a single dose of subcutaneous injection.
  Interventions: Drug: TQC2938 Injection
- TQC2938 Injection (840mg/5.6ml)-subcutaneous injection (Experimental): TQC2938 Injection is administered as a single dose of subcutaneous injection.
  Interventions: Drug: TQC2938 Injection
- TQC2938 Injection (1260mg/8.4ml) (Experimental): TQC2938 Injection is administered as a single dose of subcutaneous injection.
  Interventions: Drug: TQC2938 Injection
- TQC2938 Injection (210mg/1.4ml)-subcutaneous injection-multiple doses (Experimental): TQC2938 Injection is administered as a multiple doses of subcutaneous injection, once every 28 days, three times in total.
  Interventions: Drug: TQC2938 Injection
- TQC2938 Injection (840mg/5.6ml)-subcutaneous injection-multiple doses (Experimental): TQC2938 Injection is administered as a multiple doses of subcutaneous injection, once every 28 days, three times in total.
  Interventions: Drug: TQC2938 Injection
- TQC2938 Injection (630mg/4.2ml) (Experimental): TQC2938 Injection is administered as a multiple doses of subcutaneous injection, once every 28 days, three times in total.
  Interventions: Drug: TQC2938 Injection
- TQC2938 Placebo (Placebo Comparator): TQC2938 Placebo is administered as a single dose or multiple doses, once every 28 days, three times in total.
  Interventions: Drug: TQC2938 Placebo

INTERVENTIONS:
Drug: TQC2938 Injection — TQC2938 injection is a humanized monoclonal antibody that interfering with the signal cascade.
  Arms: TQC2938 Injection (1260mg/8.4ml); TQC2938 Injection (210mg/1.4ml)-intravenous injection; TQC2938 Injection (210mg/1.4ml)-subcutaneous injection; TQC2938 Injection (210mg/1.4ml)-subcutaneous injection-multiple doses; TQC2938 Injection (420mg/2.8ml); TQC2938 Injection (52.5mg/0.35ml); TQC2938 Injection (630mg/4.2ml); TQC2938 Injection (840mg/5.6ml)-subcutaneous injection; TQC2938 Injection (840mg/5.6ml)-subcutaneous injection-multiple doses
Drug: TQC2938 Placebo — TQC2938 Placebo is a placebo comparator
  Arms: TQC2938 Placebo

SUMMARY:
The study is designed in two phases: single-dose administration and multiple-dose administration. A randomized, double-blind, placebo-controlled trial design was used to evaluate the safety, tolerability, pharmacokinetic characteristics and immunogenicity of TQC2938 injection in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent before the study to fully understand the purpose, process and possible adverse reactions of the test.
* Adults aged between 18 and 60 years (inclusive)，both male and female;
* The male subject should weigh at least 50kg, the female subject should weigh at least 45kg. And body mass index (BMI) within 18~28 kg/m2 (inclusive);
* The subjects were able to communicate well with the investigators, voluntarily and were able to understand and follow the protocol to complete the study;
* Female patient had no plans to become pregnant for 6 months from the date of signing the informed consent to the last dose, and must use effective non-drug contraception with their sexual partners of childbearing age。

Exclusion Criteria:

* Pregnant or lactating women;
* Past medical history or current cardiac, endocrine, metabolic, renal, hepatic, gastrointestinal, skin, infection, hematological, neurological or psychiatric diseases/abnormalities, or related chronic abnormalities, or related chronic diseases, or acute diseases, and the investigator evaluated that the subject was not suitable for the trial;
* People who have abnormal and clinically significant results in vital signs, physical examination, laboratory tests, 12-lead electrocardiogram (ECG) and Chest radiograph during screening period;
* Subjects Positive for Any of Hepatitis B Virus Surface Antigen (HBsAg), Hepatitis C Virus Antibody (Anti-HCV), Human Immunodeficiency Virus Antibody (Anti-HIV), and Treponema Pallidum Antibody (Anti-TP);
* A history of clinically significant infections, including upper respiratory tract infections (URTI) and lower respiratory tract infections (LRTI), occurred within 30 days prior to and during screening and required antibiotic or antiviral treatment;
* Had undergone surgery within 8 weeks prior to screening period or expected to undergo surgery during the study period;
* Participated in any clinical trial within 3 months prior to the screening period;
* Received immunoglobulins or blood products within 30 days prior to randomization;
* Blood donation or significant blood loss of more than 400 mL within 3 months prior to randomization, or plan to donate blood within 3 months;
* Potential blood collection difficulties, can not tolerate venipuncture or have a history of fainting needles and fainting blood;
* A history of allergic reaction to treatment with another therapeutic monoclonal antibody or biologics, a history of any well-defined drug or food allergy, especially to ingredients similar to the drug in this trial;
* Those who received or planned to receive inactivated or active vaccines within 30 days prior to randomization or throughout the study period, including the follow-up period；
* Those who smoked more than 5 cigarettes/day or used a comparable amount of nicotine or nicotine-containing products in the 6 months prior to randomization, or could not stop using any tobacco products during the trial period；
* People with chronic alcohol abuse or who drank more than 14 units of alcohol per week in the 3 months prior to screening (1 unit =360 mL beer or 45 mL spirits with 40% alcohol or 150 mL wine), or who could not abstain during the test period, or who tested positive for alcohol breath；
* History of drug abuse or a positive result of urine drug test at screening;
* Received any marketed or investigational biological agent (other than vaccines) within 4 months or 5 half-lives (whichever is older) prior to randomization；
* Any prescription, over-the-counter, and herbal medicines, except vitamin products, were taken in the 4 weeks prior to randomization；
* Use of any systemic cytotoxicity or systemic immunosuppressants within 6 months prior to randomization or during the study period, or any local cytotoxin or local immunosuppressive drug within 30 days or 5 half-life periods (whichever is longer) prior to randomization or during the study period；
* Any situation in which the investigator believes that this poses a safety risk to the subject in the trial or may interfere with the conduct of the study, or that the investigator believes that the subject may not be able to complete the study or may not be able to comply with the requirements of the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | Single dose: Up to Day 113. Multiple doses: Up to Day 169
  The occurrence of all adverse events (AEs).
Serious adverse events (SAEs) | Single dose: Up to Day 113. Multiple doses: Up to Day 169
  The occurrence and incidence of all serious adverse events (SAEs).
Clinical laboratory abnormalities | Single dose: Up to Day 113. Multiple doses: Up to Day 169
  Incidence of abnormal clinical laboratory examination, vital signs, physical examination, 12-lead electrocardiogram, etc.

SECONDARY OUTCOMES:
Maximum serum concentration (Cmax) of subcutaneous injection for single dose | Single dose: pre-dose (-1 to 0 hour),1, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 264, 336, 504, 672, 1008, 1344, 1680, 2016, 2352 and 2688 hours post-dose
  The Cmax is the maximum observed serum concentration of study drug.
Maximum serum concentration (Cmax) of intravenous injection for single dose | Single dose: pre-dose (-1 to 0 hour), 0.5hours after the start of administration, and 0,0.25, 0.5, 1, 2, 4, 8, 24, 48, 72, 96, 120, 144, 168, 192, 264, 336, 504, 672, 1008, 1344, 1680, 2016, 2352, 2688 hours post-dose
  The Cmax is the maximum observed serum concentration of study drug.
Maximum serum concentration (Cmax) of subcutaneous injection for multiple doses | Multiple doses: pre-dose (-1 to 0 hour) of days 1, 29, 57, and 1, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 264, 336, 504 hours post-dose on multiple dose of days 1 and 57, and 672, 1008, 1344, 1680, 2016, 2352, 2688 hours post-dose of day 57
  The Cmax is the maximum observed serum concentration of study drug.
Time to reach maximum observed serum concentration (Tmax) of subcutaneous injection for single dose | Single dose: pre-dose (-1 to 0 hour),1, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 264, 336, 504, 672, 1008, 1344, 1680, 2016, 2352 and 2688 hours post-dose
  Time to reach maximum (peak) serum concentration following drug administration.
Time to reach maximum observed serum concentration (Tmax) of intravenous injection for single dose | Single dose: pre-dose (-1 to 0hour), 0.5hours after the start of administration, and 0,0.25, 0.5, 1, 2, 4, 8, 24, 48, 72, 96, 120, 144, 168, 192, 264, 336, 504, 672, 1008, 1344, 1680, 2016, 2352, 2688 hours post-dose
  Time to reach maximum (peak) serum concentration following drug administration.
Time to reach maximum observed serum concentration (Tmax) of subcutaneous injection for multiple doses | Multiple doses: pre-dose (-1 to 0hour) of days 1, 29, 57, and 1, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 264, 336, 504hours post-dose of days 1 and 57, and 672, 1008, 1344, 1680, 2016, 2352, 2688 hours post-dose of day 57
  Time to reach maximum (peak) serum concentration following drug administration.
Minimum concentration of drug in serum at steady state (Cmin, ss) of subcutaneous injection for multiple doses | Multiple doses: Pre-dose (-1 to 0 hour) of day 1, day 29, day 57, and 1, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 264, 336, 504 hours of day 1 and day 57, and 672, 1008, 1344, 1680, 2016, 2352, 2688 hours post-dose of day 57
  Cmin,ss is the minimum serum concentration at steady state.
Area under the concentration-time curve from 0 to last observation (AUC [0-t]) of subcutaneous injection for single dose | Single dose: pre-dose (-1 to 0 hour),1, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 264, 336, 504, 672, 1008, 1344, 1680, 2016, 2352 and 2688 hours post-dose
  Area under the concentration-time curve of the TQC2938 Injection in serum over the time interval from 0 extrapolated to the last quantifiable data point.
Area under the concentration-time curve from 0 to last observation (AUC [0-t]) of intravenous injection for single dose | Single dose: pre-dose (-1 to 0 hour), 0.5 hours after the start of administration, and 0,0.25, 0.5, 1, 2, 4, 8, 24, 48, 72, 96, 120, 144, 168, 192, 264, 336, 504, 672, 1008, 1344, 1680, 2016, 2352, 2688 hours post-dose
  Area under the concentration-time curve of the TQC2938 Injection in serum over the time interval from 0 extrapolated to the last quantifiable data point.
Area under the concentration-time curve from 0 to last observation (AUC [0-t]) of of subcutaneous injection for multiple dose | Multiple doses: pre-dose(-1 to 0 hour) of day 1, day 29, day 57, and 1, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 264, 336, 504 hours post-dose of day 1 and day 57, and 672, 1008, 1344, 1680, 2016, 2352, 2688 hours post-dose of day 57
  Area under the concentration-time curve of the TQC2938 Injection in serum over the time interval from 0 extrapolated to the last quantifiable data point.
Maximum concentration of drug in serum at steady state (Cmax, ss) of subcutaneous injection for multiple doses | Multiple doses: pre-dose (-1 to 0 hour) of day 1, day 29, day 57, and 1, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 264, 336, 504 hours post-dose of day 1 and day 57, and 672, 1008, 1344, 1680, 2016, 2352, 2688 hours post-dose of day 57
  Cmax, ss is the peak serum concentration of TQC2938 Injection during dosing interval at steady state.
Time to maximum serum concentration at steady state (Tmax, ss) of subcutaneous injection | Multiple doses: pre-dose (-1 to 0 hour) of day 1, day 29, day 57, and 1, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 264, 336, 504 hours post-dose of day 1 and day 57, and 672, 1008, 1344, 1680, 2016, 2352, 2688 hours post-dose of day 57
  Tmax,ss is defined as time to reach the peak serum concentration at steady state for TQC2938 Injection.
Area under curve of steady state (AUCss) of subcutaneous injection | Multiple doses: pre-dose (-1 to 0 hour) of day 1, day 29, day 57, and 1, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 264, 336, 504 hours post-dose of day 1 and day 57, and 672, 1008, 1344, 1680, 2016, 2352, 2688 hours post-dose of day 57
  To evaluate the pharmacokinetics (PK) of multiple ascending doses (MAD) of TQC2938 Injection in serum.
Half-life (t1/2) of subcutaneous injection for single dose | Single dose: pre-dose (-1 to 0 hour),1, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 264, 336, 504, 672, 1008, 1344, 1680, 2016, 2352 and 2688 hours post-dose
  Terminal phase elimination half-life (T1/2) is the time required for half of the drug to be eliminated from the serum.
Half-life (t1/2) of intravenous injection for single dose | Single dose: pre-dose (-1 to 0 hour), 0.5 hours after the start of administration, and 0,0.25, 0.5, 1, 2, 4, 8, 24, 48, 72, 96, 120, 144, 168, 192, 264, 336, 504, 672, 1008, 1344, 1680, 2016, 2352, 2688 hours post-dose
  Terminal phase elimination half-life (T1/2) is the time required for half of the drug to be eliminated from the serum.
Half-life (t1/2) of intravenous injection for multiple dose | Multiple doses: pre-dose (-1 to 0 hour) of day 1, day 29, day 57, and 1, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 264, 336, 504 hours post-dose of day 1 and day 57, and 672, 1008, 1344, 1680, 2016, 2352, 2688 hours post-dose of day 57
  Terminal phase elimination half-life (T1/2) is the time required for half of the drug to be eliminated from the serum.
Apparent volume of distribution (Vd/F) of subcutaneous injection for single dose | Single dose: pre-dose (-1 to 0 hour),1, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 264, 336, 504, 672, 1008, 1344, 1680, 2016, 2352 and 2688 hours post-dose
  Apparent volume of distribution of the TQC2938 Injection in serum.
Apparent volume of distribution (Vd/F) of intravenous injection for single dose | Single dose: pre-dose (-1 to 0 hour), 0.5 hours after the start of administration, and 0,0.25, 0.5, 1, 2, 4, 8, 24, 48, 72, 96, 120, 144, 168, 192, 264, 336, 504, 672, 1008, 1344, 1680, 2016, 2352, 2688 hours post-dose
  Apparent volume of distribution of the TQC2938 Injection in serum.
Apparent volume of distribution (Vd/F) of subcutaneous injection for multiple dose | Multiple doses: pre-dose (-1 to 0 hour) of day 1, day 29, day 57, and 1, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 264, 336, 504 hours post-dose of day 1 and day 57, and 672, 1008, 1344, 1680, 2016, 2352, 2688 hours post-dose of day 57
  Apparent volume of distribution of the TQC2938 Injection in serum.
Apparent clearance (CL/F) of subcutaneous injection for single dose | Single dose: pre-dose (-1 to 0 hour),1, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 264, 336, 504, 672, 1008, 1344, 1680, 2016, 2352 and 2688 hours post-dose
  Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the body.
Apparent clearance (CL/F) of intravenous injection for single dose | Single dose: pre-dose (-1 to 0 hour), 0.5 hours after the start of administration, and 0,0.25, 0.5, 1, 2, 4, 8, 24, 48, 72, 96, 120, 144, 168, 192, 264, 336, 504, 672, 1008, 1344, 1680, 2016, 2352, 2688 hours post-dose
  Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the body.
Apparent clearance (CL/F) of subcutaneous injection for multiple dose | Multiple doses: pre-dose (-1 to 0 hour) of day 1, day 29, day 57, and 1, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 264, 336, 504 hours post-dose of day 1 and day 57, and 672, 1008, 1344, 1680, 2016, 2352, 2688 hours post-dose of day 57
  Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the body.
Accumulation ratio (Rac) of subcutaneous injection for multiple dose | Multiple doses: pre-dose (-1 to 0 hour) of day 1, day 29, day 57, and 1, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 264, 336, 504 hours post-dose of day 1 and day 57, and 672, 1008, 1344, 1680, 2016, 2352, 2688 hours post-dose of day 57
  To evaluate the pharmacokinetics (PK) of multiple ascending doses (MAD) of TQC2938 Injection in serum.
Anti-drug antibodies (ADA) | Single dose: (-1 to 0 hour) (pre-dose), 672, 1344, 2016 and 2688 hours postdose. Multiple doses: (-1 to 0 hour) before the first,second and third administration, 1344 and 2688 hours after intravenous injection of Day 57
  Incidence of ADA, a participant was considered ADA-positive across the study if they had a positive reading at any time point during the study.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China